CLINICAL TRIAL: NCT00372619
Title: A Phase I/II Study of CLOLAR® (Clofarabine, IND# 73, 789) in Combination With Cytarabine in Pediatric Patients With Refractory/Relapsed Leukemia
Brief Title: Clofarabine and Cytarabine in Treating Young Patients With Refractory or Relapsed Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAML0523; CDR0000494654 (Other: Clinical Trials.gov); NCI-2009-00319 (Other: NCI Trial Identifier); COG-AAML0523 (Other: Children's Oncology Group)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-02

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; acute undifferentiated leukemia; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); childhood acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); childhood acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); childhood acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); childhood acute erythroleukemia (M6); adult acute megakaryoblastic leukemia (M7); childhood acute megakaryocytic leukemia (M7); recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Clofarabine; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Clofarabine 40 mg/m² to assess feasibility in ALL patients. (Experimental): Clofarabine 40 mg/m² to assess feasibility in ALL patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 40 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: methotrexate; Other: laboratory biomarker analysis
- Clofarabine 40 mg/m² to assess feasibility in AML patients. (Experimental): Clofarabine 40 mg/m² to assess feasibility in AML patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 40 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: methotrexate; Other: laboratory biomarker analysis
- Clofarabine 52 mg/m² to assess feasibility in ALL patients. (Experimental): Clofarabine 52 mg/m² to assess feasibility in ALL patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: methotrexate; Other: laboratory biomarker analysis
- Clofarabine 52 mg/m² to assess efficacy in ALL patients. (Experimental): Clofarabine 52 mg/m² to assess efficacy in ALL patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: methotrexate; Other: laboratory biomarker analysis
- Clofarabine 52 mg/m² to assess feasibility in AML patients. (Experimental): Clofarabine 52 mg/m² to assess feasibility in AML patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: methotrexate; Other: laboratory biomarker analysis
- Clofarabine 52 mg/m² to assess efficacy in AML patients (Experimental): Clofarabine 52 mg/m² to assess efficacy in AML patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: methotrexate; Other: laboratory biomarker analysis
- Clofarabine 52 mg/m² to assess efficacy - ambiguous lineage pt (Experimental): Clofarabine 52 mg/m² to assess efficacy in acute leukemia of ambiguous lineage patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: methotrexate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: clofarabine — Given IV for 5 days
  Other Names: Cl-F-Ara-A; CAFdA; 2-Chloro-9-(2-deoxy-2-fluoro-beta-D-arabinofuranosyl)-9H-purin-6-amine; Clolar; Evoltra; NSC# 606,869; IND # 73,789
Drug: cytarabine — Given IV
  Other Names: Cytosine arabinoside; Ara-C; Cytosar; NSC #063878
Drug: methotrexate — Given intrathecally or IT age based dosage
  Other Names: MTX; amethopterin; Trexall; NSC #000740
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of clofarabine when given together with cytarabine and to see how well they work in treating young patients with refractory or relapsed acute myeloid leukemia or acute lymphoblastic leukemia. (Phase I closed to enrollment as of 09/16/09)

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define the overall response rate (complete remission or remission without platelet recovery) in young patients with relapsed or refractory acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) treated with clofarabine in combination with cytarabine.

Secondary

* To determine the safety profile and tolerability of clofarabine when given in combination with cytarabine in patients with and without prior stem cell transplantation.
* To identify apoptosis specific genes that are important in mediating response to clofarabine and cytarabine.
* To quantitate the level of human equilibrative nucleoside transporter proteins (hENT1 and hENT2) and human concentrative nucleoside transporter proteins (hCNT2 and hCNT3) in blasts of these patients.
* To determine gene expression profiles at study entry and at time of relapse in order to isolate profiles that may predict response and also to complement apoptosis specific protein arrays.
* To perform serial measurements of minimal residual disease (MRD) to provide an objective determination of the effectiveness of this treatment regimen and to correlate with post remission events (relapse, death).
* To perform FLT3/ITD analysis to help determine the prevalence and clinical significance of this somatic mutation in patients with relapsed AML.

OUTLINE: This is a multicenter, phase I, dose-escalation study of clofarabine followed by a phase II study. Patients are stratified according to disease (acute lymphoblastic leukemia [ALL] vs acute myeloid leukemia [AML]). (Phase I closed to accrual as of 09/16/09)

* Intrathecal CNS prophylaxis (all patients with ALL and at physician's discretion for patients with AML or acute leukemia of ambiguous lineage): Patients receive intrathecal (IT) cytarabine on day 0 of the first course of induction therapy. Patients also receive IT methotrexate on day 1 of the second course of induction therapy and on day 1 of all courses of maintenance therapy.
* Induction therapy:

  * Course 1: Patients receive cytarabine IV over 2 hours and clofarabine IV over 2 hours on days 1-5. Patients with ≥ 5% blasts (i.e., M2 or M3 bone marrow) at days 14-21 proceed immediately to course 2 of induction therapy. Patients with < 5% blasts (i.e., M1 bone marrow) may proceed to course 2 of induction therapy at blood count recovery or at day 42.
  * Course 2: Patients receive clofarabine IV over 2 hours followed by cytarabine IV over 2 hours on days 1-5. After the second course of induction therapy, patients with M2 or M3 bone marrow at days 14-21 are removed from the study. Patients with M1 bone marrow proceed to maintenance therapy 14-42 days after the initiation of course 2.
* Maintenance therapy: Patients receive clofarabine and cytarabine as in induction therapy. Treatment repeats every 14-42 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood and bone marrow sample collection periodically for correlative laboratory studies.

After completion of study therapy, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 87 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML) with ≥ 5% blasts in the bone marrow (M2/M3 bone marrow) with or without extramedullary disease
  * Acute lymphoblastic leukemia (ALL) with > 25% blasts in the bone marrow (M3 bone marrow) with or without extramedullary disease
  * Acute leukemia of ambiguous lineage with ≥ 5% blasts in the bone marrow (M2/M3 bone marrow) with or without extramedullary disease
* Disease must have relapsed after or be refractory to prior induction therapy

  * Patients with AML or acute leukemia of ambiguous lineage must be in first relapse OR refractory to first induction therapy with ≤ 1 attempt at remission induction

    * Patients with AML who enroll on the phase I portion of the study must have received prior mitoxantrone hydrochloride and cytarabine for newly diagnosed AML (phase I closed to accrual as of 09/16/09)
  * Patients with ALL must be in second or third relapse (≤ 3 prior induction regimens) OR refractory to reinduction in first relapse

    * Patients with ALL refractory to first induction therapy are not eligible
* No acute promyelocytic leukemia
* No CNS 3 involvement (i.e., WBC ≥ 5/μL in the cerebrospinal fluid with blasts present on cytospin)

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (> 16 years of age) OR Lansky PS 50-100% (≤ 16 years of age) OR ECOG PS 0-2
* Life expectancy ≥ 8 weeks
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min
* Direct bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 2.5 times ULN (unless it is related to leukemic involvement)
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 45% by gated radionuclide study
* No evidence of dyspnea at rest or exercise intolerance
* Pulse oximetry > 94% at room air
* Amylase ≤ 1.5 times ULN
* Lipase < 1.5 times ULN
* No active, uncontrolled grade 3 or 4 infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No known hepatitis B or C infection or history of cirrhosis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy*
* At least 14 days since prior cytotoxic therapy (except hydroxyurea and intrathecal chemotherapy)*
* At least 7 days since prior biologic agent*
* At least 14 days since prior monoclonal antibody therapy*
* No more than 1 prior autologous or allogeneic hematopoietic stem cell transplantation

  * No evidence of active graft-vs-host disease
  * At least 4 months since transplantation
* No other concurrent chemotherapy or immunomodulating agents
* No other concurrent investigational therapy NOTE: *Patients who relapse during ALL maintenance therapy do not require a waiting period.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2007-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bassem I. Razzouk, MD, Study Chair — St. Vincent Indianapolis Hospital; Todd Cooper, DO, Study Chair — University of Alabama at Birmingham
Locations (79):
- United States (74):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Southern California Permanente Medical Group, Downey, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Colorado Center for Cancer and Blood Disorders, Aurora, Colorado
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients.: Clofarabine 40 mg/m² to assess feasibility in ALL patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 40 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  clofarabine: Given IV for 5 days
  cytarabine: Given IV
  methotrexate: Given intrathecally or IT age based dosage
  laboratory biomarker analysis
- Clofarabine 40 mg/m² to Assess Feasibility in AML Patients.: Clofarabine 40 mg/m² to assess feasibility in AML patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 40 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 40 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  clofarabine: Given IV for 5 days
  cytarabine: Given IV
  methotrexate: Given intrathecally or IT age based dosage
  laboratory biomarker analysis
- Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients.: Clofarabine 52 mg/m² to assess feasibility in ALL patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  clofarabine: Given IV for 5 days
  cytarabine: Given IV
  methotrexate: Given intrathecally or IT age based dosage
  laboratory biomarker analysis
- Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients.: Clofarabine 52 mg/m² to assess efficacy in ALL patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  clofarabine: Given IV for 5 days
  cytarabine: Given IV
  methotrexate: Given intrathecally or IT age based dosage
  laboratory biomarker analysis
- Clofarabine 52 mg/m² to Assess Feasibility in AML Patients.: Clofarabine 52 mg/m² to assess feasibility in AML patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  clofarabine: Given IV for 5 days
  cytarabine: Given IV
  methotrexate: Given intrathecally or IT age based dosage
  laboratory biomarker analysis
- Clofarabine 52 mg/m² to Assess Efficacy in AML Patients: Clofarabine 52 mg/m² to assess efficacy in AML patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  clofarabine: Given IV for 5 days
  cytarabine: Given IV
  methotrexate: Given intrathecally or IT age based dosage
  laboratory biomarker analysis
- Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt: Clofarabine 52 mg/m² to assess efficacy in acute leukemia of ambiguous lineage patients. Patients receive Cycle 1 (14-42 days) Cytarabine IT (aged based dosage 1-1.99 30 mg, 2-2.99 50 mg, ≥ 3 years 70 mg on Day 0, Clofarabine IV (dosage 52 mg/m2/dose) on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Cycle 2 (14-42 days) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5. Maintenance cycles 1-10 (14-42 days each) Methotrexate IT (age based dosage 1-1.99 8 mg, 2-2.99 10 mg, ≥ 3 12 mg) on day 1, Clofarabine IV 52 mg/m2/dose on days 1-5, and High Dose Cytarabine IV 1000 mg/m2/dose on days 1-5.
  clofarabine: Given IV for 5 days
  cytarabine: Given IV
  methotrexate: Given intrathecally or IT age based dosage
  laboratory biomarker analysis
Period: Overall Study
Arm/Group | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt
Started | 8 | 2 | 3 | 10 | 7 | 42 | 2
Completed | 8 | 2 | 3 | 10 | 7 | 39 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Ineligible | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Inevaluable | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt | Total
Number analyzed (Participants) | 8 | 2 | 3 | 10 | 7 | 42 | 2 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 1 | 3 | 9 | 7 | 34 | 1 | 62
  Between 18 and 65 years | 1 | 1 | 0 | 1 | 0 | 8 | 1 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.75 (6.37) | 15.09 (6.33) | 13.09 (1.54) | 9.16 (6.69) | 9.01 (5.79) | 12.01 (7.12) | 19.65 (1.80) | 15.13 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 2 | 4 | 3 | 20 | 1 | 35
  Male | 3 | 2 | 1 | 6 | 4 | 22 | 1 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 0 | 7 | 0 | 11
  Not Hispanic or Latino | 6 | 2 | 0 | 8 | 6 | 35 | 2 | 59
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 8 | 0 | 11
  White | 6 | 1 | 2 | 8 | 7 | 28 | 2 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 4 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 1 | 3 | 8 | 7 | 37 | 2 | 65
  Canada | 1 | 1 | 0 | 2 | 0 | 5 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (CR for ALL Patients), (CR + CRp for AML Patients)
Description: Overall response for ALL patients: CR - complete remission (attainment of an M1 bone marrow (< 5% blasts) with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral counts (absolute neutrophil count (ANC) > 750/μL and platelet count > 75,000/μL).
  Overall response for AML patients: (CR + CRp), defined as:
  CR - complete remission (attainment of an M1 bone marrow (<5% blasts) with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral blood counts (absolute neutrophil count (ANC) > 1000/uL and platelet count > 100,000/uL)) or CRp - remission without platelet recovery (Attainment of an M1 bone marrow (<5% blasts) with no evidence of circulating blasts or extramedullary disease and with recovery of absolute neutrophil count (ANC) > 1000/uL and platelet transfusion independence (defined as: no platelet transfusions x 1 week)).
Time Frame: 2 cycles or up to 84 days
Measure: Number; unit: participants
Arm/Group | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt
Number analyzed (Participants) | 8 | 2 | 3 | 10 | 7 | 39 | 2
participants | 1 | 2 | 0 | 2 | 2 | 19 | 2

2. Secondary Outcome: Safety and Tolerability as Measured by CTCAE v3.0
Description: Number of participants with at least one grade 3 or higher adverse event during therapy.
Time Frame: End of therapy
Population: Ineligible (n=2) and inevaluable (n=1) patients are excluded
Measure: Number; unit: number participants
Arm/Group | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt
Number analyzed (Participants) | 8 | 2 | 3 | 10 | 7 | 39 | 2
number participants | 7 | 2 | 3 | 10 | 7 | 35 | 2

3. Secondary Outcome: Correlate the Expression of Apoptosis Specific Genes
Description: Correlate the expression of apoptosis specific genes with chemoresistance and determine whether therapy with clofarabine is able to overcome blocks in apoptosis through modulation of gene expression. Gene expression analysis will be performed on specimens obtained during therapy. Apoptosis specific microarray data will be analyzed using GeneTraffic software (Iobion Informatics, La Jolla CA).
Time Frame: End of therapy
Population: The analysis was not completed, because the tissue microarray was unsuccessful.
Arm/Group | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: There are n=42 pts enrolled to group Clofarabine 52 mg/m² to Assess Efficacy in AML Patients, 2 pts ineligible & 1 inevaluable for response. For toxicity, ineligible pts are excluded, but the inevaluable pt is included for analysis of toxicity resulting in n=40. OM #2 reports the number of pts having at least 1, gr 3 or higher AE during therapy. Pts with SAEs are not determined by this definition, but by whether a pt had at least 1 reportable AE requiring an AdEERs report during therapy.
Arm/Group | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt
Serious Adverse Events (participants affected / at risk) | 5/8 | 2/2 | 2/3 | 7/10 | 3/7 | 14/40 | 2/2
Other Adverse Events (participants affected / at risk) | 8/8 | 2/2 | 3/3 | 10/10 | 7/7 | 38/40 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. (N=8) | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. (N=2) | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. (N=3) | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. (N=10) | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. (N=7) | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients (N=40) | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt (N=2)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 1 | 6 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 4 | 0 | 1 | 3 | 2 | 8 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine 40 mg/m² to Assess Feasibility in ALL Patients. (N=8) | Clofarabine 40 mg/m² to Assess Feasibility in AML Patients. (N=2) | Clofarabine 52 mg/m² to Assess Feasibility in ALL Patients. (N=3) | Clofarabine 52 mg/m² to Assess Efficacy in ALL Patients. (N=10) | Clofarabine 52 mg/m² to Assess Feasibility in AML Patients. (N=7) | Clofarabine 52 mg/m² to Assess Efficacy in AML Patients (N=40) | Clofarabine 52 mg/m² to Assess Efficacy - Ambiguous Lineage pt (N=2)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 1 | 3 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 1 | 4 | 1 | 14 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 5 | 3 | 11 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2 | 5 | 1 | 10 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0 | 5 | 0 | 6 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Creatinine increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 4 | 10 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 1 | 1 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 5 | 4 | 12 | 0
Fever (General disorders) | 1 | 0 | 1 | 3 | 1 | 5 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
GGT increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 7 | 0
Gum infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 3 | 0 | 2 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 5 | 1 | 7 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 6 | 3 | 9 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 4 | 0 | 5 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3 | 1 | 7 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 3 | 13 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 2 | 4 | 1
Hypotension (Vascular disorders) | 2 | 0 | 1 | 0 | 1 | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 2 | 1 | 2 | 4 | 17 | 1
INR increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 4 | 4 | 10 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 2 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 3 | 0 | 0 | 2 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 3 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 5 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 4 | 5 | 9 | 1
Watering eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
White blood cell decreased (Investigations) | 2 | 0 | 0 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.